CLINICAL TRIAL: NCT06537479
Title: Combined Effects of Buteyko Breathing Technique and Chest Wall Mobilization on Pulmonary Functions and Quality of Life in Chronic Smokers
Brief Title: Combined Effects of Buteyko Breathing Technique and Chest Wall Mobilization on Pulmonary Functions and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0373
Record Dates: First submitted 2024-06-24; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Chronic Smokers
Keywords: Buteyko Breathing Technique, Chest wall Mobilization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko breathing technique, Chest wall mobilization (Experimental): Deep breathing exercises for 5 minutes. After the 5-minute resting interval Buteyko breathing technique and chest wall mobilization of 5 minutes Chest wall mobilization with 8-10 repetitions. Total time duration will be 30 minutes. 2 sessions per week
  Interventions: Other: Buteyko breathing technique; Other: Chest Wall Mobilization
- Buteyko breathing technique (Active Comparator): Deep breathing for 5 minutes as a baseline Buteyko technique of 2 sets of 8-10 repetitions for 2 days a week. Chest wall mobilization will not be included in Group 2. Repeat the breathing cycle for 5-10 minutes, 2-3 times a day. Total time duration will be 30 minutes.
  Interventions: Other: Buteyko breathing technique

INTERVENTIONS:
Other: Buteyko breathing technique — Participants will be advised to sit in a comfortable and relaxed position and take a shallow breath through nose, partially filling the lungs. Hold breath for 2-3 seconds and exhale slowly through the nose and emptying the lungs.
Other: Chest Wall Mobilization — It started with positioning, sitting or standing with good posture, and relaxing shoulders and arms. Hands were placed on the chest with fingers wide and thumbs on side of ribcage. Inhale deep breaths with expansion of chest and hands move outward. Exhale slowly allowed the chest to drop and the hands to move inward.
  Arms: Buteyko breathing technique, Chest wall mobilization

SUMMARY:
The study aims to evaluate the effects of Buteyko breathing techniques with and without chest wall mobilization on pulmonary functions, and quality of life in chronic smokers. The study design will be a randomized clinical trial. The study will be completed in 10 months after the approval of the synopsis from the Ethical Committee of RCRS & AHS. A non-probability convenient sampling technique will be used to recruit the individuals. Group 1-Buteyko breathing technique + Chest Wall Mobilization and Group 2-Buteyko Breathing Technique + Without Chest Wall Mobilization

DETAILED DESCRIPTION:
This randomized clinical trial will evaluate the combined effect of the Buteyko breathing technique and chest wall mobilization on pulmonary functions and quality of life in chronic smokers. A sample size of 40 is calculated through a non-probability convenient sampling technique. Participants will be recruited into Group 1 and Group 2 by lottery method (without replacement). Group 1 will be engaged in the Buteyko breathing technique + Chest Wall Mobilization and Group 2 will undergo Buteyko Breathing Technique + Without Chest Wall Mobilization. Pre and post-outcome measures of pulmonary functions will be measured through a digital spirometer and quality of life will be assessed by the St George Quality of Life Questionnaire.

Spirometry assesses the amount and speed of air that can be inhaled and exhaled. Key measurements include Forced Vital Capacity (FVC): The maximum volume of air forcefully exhaled after a full inhalation. Forced Expiratory Volume in 1 Second (FEV1): The volume of air exhaled in the first second of the FVC test, indicates how quickly the lungs can be emptied.

St Saint Georg quality of life questionnaire for assessing the QOL. The SGRQ is a standardized self-administered airway disease-specific questionnaire divided into 2 subscales, a total of 12 questions. For each subscale and the overall questionnaire, scores range from zero (no impairment) to 100 (maximum impairment).

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants were included
* The age of participants was 40 -55 years.
* Individuals who fulfilled the criteria of smoking which is calculated by multiplying the number of packs smoked per day by the number of years smoked were included.
* Individuals who are current smokers or history of long-term smoking were included.
* Predicted values FEV1 < 75% and FEV1/FVC <70%

Exclusion Criteria:

* Participants with neurological disorders were excluded
* Participants with musculoskeletal disorders were excluded as it affects the physical activity of the 6-minute walk test.
* Participants having any pulmonary complications or lung disease were excluded.
* Participants previously involved in any other exercise or physical activity were excluded.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-08-13 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
FEV1(Forced Expiratory Volume per second) | Pre and Post after 1 week
  Pulmonary Function Test using Digital Spirometer. • Forced Vital Capacity (FVC): the amount of air that can be forcefully exhaled after taking a complete breath.
FVC(Forced Vital Capacity) | Pre and Post after 1 week
  Pulmonary Function Test using Digital Spirometer. the amount of air expelled during the first second of the forced ventilation test (FVC), which measures how rapidly the lungs can empty.
St George Questionnaire | Pre and Post after 1 week
  To assess the Quality of Life. The total questionnaire score is 100 (highest impairment) while the subscale values range from zero (no impairment)

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem Shehzadi, Mphil, Principal Investigator — Riphah International University
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No